CLINICAL TRIAL: NCT04382794
Title: Sitagliptin Treatment in Diabetic COVID-19 Positive Patients: Retrospective Study
Brief Title: Sitagliptin Treatment in Diabetic COVID-19 Positive Patients
Acronym: SIDIACO-RETRO'
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: Papa Giovanni XXIII Hospital (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Humanitas Hospital, Italy (Other); Ospedale dell'Angelo, Venezia-Mestre (Other); University of Pavia (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Clinical Professor, University of Milan
Other Study IDs: 5/2020
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Covid19
Keywords: Covid19; Sitagliptin; Diabetes Mellitus, Type 2
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- DMT2 COVID19 positive patients treated with Sitagliptin: The anonymous data relating to the clinical, laboratory and instrumental parameters of patients hospitalized for COVID-19 and suffering from type 2 diabetes treated with Sitagliptin will be extracted from the medical records currently in use in the centers participating in the study. The data will be anonymous and not attributable to individual subjects
  Interventions: Drug: Retrospective case-control analysis
- DMT2 COVID19 positive patients not treated with Sitagliptin: The anonymous data relating to the clinical, laboratory and instrumental parameters of patients hospitalized for COVID-19 and suffering from type 2 diabetes not treated with Sitagliptin will be extracted from the medical records currently in use in the centers participating in the study. The data will be anonymous and not attributable to individual subjects
  Interventions: Drug: Retrospective case-control analysis

INTERVENTIONS:
Drug: Retrospective case-control analysis — Evaluation of clinical, laboratory and instrumental parameters of diabetic patients during hospitalization for COVID-19. The data will be extracted anonymously from the computerized medical records commonly used in clinical practice by the centers involved in the study

SUMMARY:
Coronavirus Pathology is frequently associated with both diabetes mellitus and metabolic syndrome. In particular, results of observational studies and meta-analyzes configure diabetes as one of the main risk factors for the development of complications and unfavorable course of SARS (Severe Acute Respiratory Syndrome) and MERS (Middle East Respiratory Syndrome), the syndromes caused respectively by SARS- VOC coronavirus and MERS-COV coronavirus. The available data confirm this association also in the clinical picture of the infection supported by SARS-COV 2 (COVID-19). In the epidemic outbreak that erupted at the beginning of 2020 in the Lombardy Region, about two thirds of the patients who died from COVID-19 were affected by diabetes mellitus. COVID-19 occurs in 70% of cases with an inflammatory pathology of the airways that can be fed by a cytokine storm and result in severe respiratory failure (10% cases) and death (5%). At the moment, the mainly involved pathophysiological molecular mechanisms are not clearly defined. It has been hypothesized that the transmembrane glycoprotein type II CD26, known for the enzyme activity Dipeptilpeptidase 4 exerted by its extracellular domain, may play a fundamental role in this process. In addition, it is considerably expressed at the parenchyma and lung interstitium level and carries out both systemic and paracrine enzymatic activity, modulating the activity of various proinflammatory cytokines, growth factors and vasoactive peptides at the level of the deep respiratory tract. The pulmonary parenchyma and the interstitium express significantly the Dipeptilpeptidase 4 protein, which in the Middle East Respiratory Syndrome favors the entry of the virus into the cells, thus allowing the virus to replicate within the cells and thus spread throughout the cell inside the organism. Dipeptilpeptidase 4 regulates the function of bioactive peptides and above all of cytokines, vasoactive peptides and chemokines present at the level of the mesothelium, of the deep respiratory tract (alveolar epithelium and alveolar bronchus), of endothelial and immune cells triggering the inflammatory storm. In line with this evidence, it has been hypothesized that acute respiratory disease from Coronavirus may depend on the massive localization of Dipeptilpeptidase 4 in lung tissue. Furthermore, the involvement of Dipeptilpeptidase 4 in other chronic respiratory diseases has been demonstrated. Starting from these observations we hypothesized that the selective blockade of Dipeptilpeptidase 4 can favorably modulate the pulmonary inflammatory response in the subject affected by COVID-19. Among the drugs that selectively block Dipeptilpeptidase 4, the one with greater affinity precisely for Dipeptilpeptidase 4 is Sitagliptin.

DETAILED DESCRIPTION:
An observational, retrospective-case control, multi-center study is proposed to evaluate any effects of Sitagliptin on clinical, laboratory and instrumental parameters in the course of hospitalization for COVID-19. The data will be extracted anonymously from the computerized medical records commonly used in clinical practice by the centers involved in the study. The evaluation will be performed by comparing the parameters of COVID-19 positive diabetic patients treated with Sitagliptin with those of a group of COVID-19 positive diabetic patients not treated with Sitagliptin. All diabetic subjects treated with Sitagliptin (100 mg / day, 50 mg / day or 25 mg / day) and all diabetic subjects not treated with Sitagliptin, eligible for inclusion / exclusion criteria, will be included in the analysis.

The clinical data of patients that will be collected anonymously during hospitalization will include: smoking habit, remote medical history aimed at assessing the presence of comorbidities (atrial fibrillation, heart failure, hypertension, arterial hypertension, chronic obstructive pulmonary disease, other lung disease, chronic renal failure, decay cognitive, Parkinson's disease, autoimmune diseases), pharmacological history (treatment introduced during hospitalization for COVID-19, respiratory failure or other complications; use of ACE-inhibitors, sartans, calcium channel blockers, diuretics, antiarrhythmics, beta blockers, anti-aggregants, anticoagulants, neuroleptics ). Anthropometric parameters including blood pressure measurement and BMI will also be collected.

For all patients, the following data will be collected at the baseline (first data available upon entry into the hospitalization regime) and upon discharge:

* Clinical picture and symptoms (presence of cough, body temperature, respiratory rate, need for ventilatory support, duration of ventilatory support in days, duration of oxygen therapy in day, duration of hospitalization in Intensive Care Unit in days, total length of stay in days, blood gas parameters, PaO2 / FiO2 ratio, oxygen saturation by pulse oximeter)
* Routine blood chemistry tests performed in hospitalization (e.g. glycemia, reactive protein C, blood count with formula, erythrocyte sedimentation rate, blood gas analysis, LDH, inflammation indices).
* Instrumental exams (chest x-ray)
* glycated hemoglobin
* Serum creatinine and Estimated Glomerular Filtration Rate (estimated with CKD-EPI)
* Presence of specific comorbidities for diabetes
* Average daily blood sugar levels (from capillary blood)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes, according to ADA 2020 criteria
* Diagnosis of COVID-19 (positive SARS-COV2 RNA buffer) with pneumonia, with or without an increase in inflammation indexes, with or without respiratory failure

Exclusion Criteria:

* Pregnancy
* Type 1 diabetes
* Presence of other acute infections in place
* Presence of serious diseases or conditions that make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The anonymous data of diabetic patients hospitalized for COVID19 in the hospitals participating in the study will be collected
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Clinical parameter of acute lung disease | 1 month
  Clinical evaluation of physiological parameter "cough" associated with acute lung disease from the beginning of the study to the end of the study
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "oxygen saturation by the use of a pulse oximeter" of acute lung disease from the beginning of the study to the end of the study
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "body temperature" of acute lung disease from the beginning of the study to the end of the study
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "PaO2/FiO2" of acute lung disease from the beginning of the study to the end of the study
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "respiratory rate" of acute lung disease from the beginning of the study to the end of the study
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "need for ventilator support" of acute lung disease from the beginning of the study to the end of the study
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "duration in days of ventilator support, duration in days of oxygen therapy, duration in days of hospitalization, duration in days in the Intensive Care Unit, total length of stay in hospital" of acute lung disease from the beginning of the study to the end of the study
Death | 1 month
  Death of the patient during hospitalization due to COVID19

SECONDARY OUTCOMES:
Biochemical parameter of acute lung disease | 1 month
  Variation of the biochemical parameter "reactive C protein" of acute lung disease from the beginning of the study to the end of the study
Biochemical parameter of acute lung disease | 1 month
  Variation of the biochemical parameter "blood count with formula" of acute lung disease from the beginning of the study to the end of the study
Biochemical parameter of acute lung disease | 1 month
  Variation of the biochemical parameter "erythrocyte sedimentation rate" of acute lung disease from the beginning of the study to the end of the study
Biochemical parameter of acute lung disease | 1 month
  Variation of the biochemical parameter "blood gas analysis" of acute lung disease from the beginning of the study to the end of the study
Biochemical parameter of acute lung disease | 1 month
  Variation of the biochemical parameter "LDH" of acute lung disease from the beginning of the study to the end of the study
Biochemical parameter of acute lung disease | 1 month
  Variation of the biochemical parameter "fasting blood glucose" of acute lung disease from the beginning of the study to the end of the study
Clinical parameter of acute lung disease | 1 month
  Variation of the clinical parameter "chest X ray" of acute lung disease from the beginning of the study to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD, PhD, Principal Investigator — ASST FBF Sacco
Locations (6):
- Italy (6):
  - ASST FBF-Sacco P.O. Sacco, Milan, MI
  - Papa Giovanni XXIII Hospital, Bergamo
  - Ospedale dell'Angelo, Venezia-Mestre, Mestre
  - Humanitas Hospital, Milan
  - University of Pavia, Pavia
  - IRCCS Policlinico S. Matteo, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang JK, Feng Y, Yuan MY, Yuan SY, Fu HJ, Wu BY, Sun GZ, Yang GR, Zhang XL, Wang L, Xu X, Xu XP, Chan JC. Plasma glucose levels and diabetes are independent predictors for mortality and morbidity in patients with SARS. Diabet Med. 2006 Jun;23(6):623-8. doi: 10.1111/j.1464-5491.2006.01861.x. PMID 16759303
- [Background] Perlman S, Azhar EI, Memish ZA, Hui DS, Zumla A. Confronting the persisting threat of the Middle East respiratory syndrome to global health security. Lancet Infect Dis. 2020 Feb;20(2):158-160. doi: 10.1016/S1473-3099(19)30347-0. Epub 2019 Jul 3. No abstract available. PMID 31279728
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Zou H, Zhu N, Li S. The emerging role of dipeptidyl-peptidase-4 as a therapeutic target in lung disease. Expert Opin Ther Targets. 2020 Feb;24(2):147-153. doi: 10.1080/14728222.2020.1721468. Epub 2020 Jan 31. PMID 31971463
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Meyerholz DK, Lambertz AM, McCray PB Jr. Dipeptidyl Peptidase 4 Distribution in the Human Respiratory Tract: Implications for the Middle East Respiratory Syndrome. Am J Pathol. 2016 Jan;186(1):78-86. doi: 10.1016/j.ajpath.2015.09.014. Epub 2015 Nov 18. PMID 26597880
- [Background] Lambeir AM, Durinx C, Scharpe S, De Meester I. Dipeptidyl-peptidase IV from bench to bedside: an update on structural properties, functions, and clinical aspects of the enzyme DPP IV. Crit Rev Clin Lab Sci. 2003 Jun;40(3):209-94. doi: 10.1080/713609354. PMID 12892317
- [Background] Schade J, Stephan M, Schmiedl A, Wagner L, Niestroj AJ, Demuth HU, Frerker N, Klemann C, Raber KA, Pabst R, von Horsten S. Regulation of expression and function of dipeptidyl peptidase 4 (DP4), DP8/9, and DP10 in allergic responses of the lung in rats. J Histochem Cytochem. 2008 Feb;56(2):147-55. doi: 10.1369/jhc.7A7319.2007. Epub 2007 Oct 29. PMID 17967935
- [Derived] Bolla AM, Loretelli C, Montefusco L, Finzi G, Abdi R, Ben Nasr M, Lunati ME, Pastore I, Bonventre JV, Nebuloni M, Rusconi S, Santus P, Zuccotti G, Galli M, D'Addio F, Fiorina P. Inflammation and vascular dysfunction: The negative synergistic combination of diabetes and COVID-19. Diabetes Metab Res Rev. 2022 Oct;38(7):e3565. doi: 10.1002/dmrr.3565. Epub 2022 Jul 22. PMID 35830597